CLINICAL TRIAL: NCT00252733
Title: Effects of Candesartan Cilexetil (Candesartan) on Diabetic Retinopathy in Type 1 Diabetic Patients Without Retinopathy.
Brief Title: Diabetic Retinopathy Candesartan Trials
Acronym: DIRECT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D2453C00045; DIRECT; SH-AHM-0045
Record Dates: First submitted 2005-11-10; First posted 2005-11-15 (Estimated); Results first posted 2012-04-13 (Estimated); Last update posted 2014-05-14 (Estimated); Status verified 2014-04

CONDITIONS: Type 1 Diabetes
Keywords: Diabetes Mellitus, Insulin-Dependent
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — candesartan cilexetil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (No Intervention): Placebo
- 2 (Experimental): candesartan cilexetil
  Interventions: Drug: candesartan cilexetil

INTERVENTIONS:
Drug: candesartan cilexetil — 32 mg once daily oral tablet given over 60 months
  Other Names: ATACAND
  Arms: 2

SUMMARY:
The primary objective is to determine whether candesartan, compared to placebo reduces the incidence of diabetic retinopathy in normotensive, normoalbuminuric type 1 diabetic patients without retinopathy.

The secondary objective is to determine whether candesartan, compared to placebo, beneficially influences the rate of change in urinary albumin excretion rate (UAER).

This study is part of the DIRECT Programme also including secondary prevention studies of diabetic retinopathy in both type 1 and type 2 diabetes. The primary objective for all three pooled studies is to determine whether candesartan, compared to placebo, reduces the incidence of microalbuminuria in type 1 and type 2 diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes diagnosed before age of 36 years and in need for continuous insulin treatment within 1 year of diagnosis of diabetes are included.
* Duration of diabetes for > 1 year and < 15 years with stable diabetic therapy within last 6 months.
* Patients with untreated resting mean sitting SBP < 130 mmHg, mean sitting DBP < 85 mmHg and with retinal photograph grading level 10/10 (on ETDRS severity scale).

Exclusion Criteria:

* Patients with the following conditions are excluded from participation in the study:
* Cataract or media opacity of a degree which precludes taking gradable retinal photographs
* Angle closure glaucoma, which precludes pharmacological dilatation of the pupil
* History of retinopathy
* History or presence of clinical significant macular oedema (CSME)
* History or evidence of photocoagulation of the retina Other retinal conditions which may mask assessment, eg, retinal vein occlusion
* Positive micral dipstick test
* Presence of secondary diabetes
* Pregnant or lactating women or women of child bearing potential not practicing an adequate method of contraception
* Need of treatment with ACE-inhibitor
* Haemodynamically significant aortic or mitral valve stenosis
* Known renal artery stenosis or kidney transplantation
* Hypersensitivity to study drug
* Severe concomitant disease which may interfere with the assessment of the patient, eg, malignancy, as judged by the investigator

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5238 (Actual)
Dates: Start 2001-06; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Atacand Medical Science Director, MD, Study Director — AstraZeneca
Locations (3):
- Australia (2):
  - Research Site, Herston
  - Research Site, Perth
- Research Site, Odense, Denmark

REFERENCES:
- [Derived] Natale P, Palmer SC, Navaneethan SD, Craig JC, Strippoli GF. Angiotensin-converting-enzyme inhibitors and angiotensin receptor blockers for preventing the progression of diabetic kidney disease. Cochrane Database Syst Rev. 2024 Apr 29;4(4):CD006257. doi: 10.1002/14651858.CD006257.pub2. PMID 38682786
- [Derived] Sjolie AK, Klein R, Porta M, Orchard T, Fuller J, Parving HH, Bilous R, Aldington S, Chaturvedi N. Retinal microaneurysm count predicts progression and regression of diabetic retinopathy. Post-hoc results from the DIRECT Programme. Diabet Med. 2011 Mar;28(3):345-51. doi: 10.1111/j.1464-5491.2010.03210.x. PMID 21309844
- [Derived] Porta M, Hainer JW, Jansson SO, Malm A, Bilous R, Chaturvedi N, Fuller JH, Klein R, Orchard T, Parving HH, Sjolie AK; DIRECT Study Group. Exposure to candesartan during the first trimester of pregnancy in type 1 diabetes: experience from the placebo-controlled DIabetic REtinopathy Candesartan Trials. Diabetologia. 2011 Jun;54(6):1298-303. doi: 10.1007/s00125-010-2040-1. Epub 2011 Jan 12. PMID 21225239
- [Derived] Bilous R, Chaturvedi N, Sjolie AK, Fuller J, Klein R, Orchard T, Porta M, Parving HH. Effect of candesartan on microalbuminuria and albumin excretion rate in diabetes: three randomized trials. Ann Intern Med. 2009 Jul 7;151(1):11-20, W3-4. doi: 10.7326/0003-4819-151-1-200907070-00120. Epub 2009 May 18. PMID 19451554
- [Derived] Chaturvedi N, Porta M, Klein R, Orchard T, Fuller J, Parving HH, Bilous R, Sjolie AK; DIRECT Programme Study Group. Effect of candesartan on prevention (DIRECT-Prevent 1) and progression (DIRECT-Protect 1) of retinopathy in type 1 diabetes: randomised, placebo-controlled trials. Lancet. 2008 Oct 18;372(9647):1394-402. doi: 10.1016/S0140-6736(08)61412-9. Epub 2008 Sep 25. PMID 18823656
- See also: Related Info — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=308&filename=CSR-D2453C00045.pdf
- See also: CSR-D2453C00045.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=308&filename=CSR-D2453C00045.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First subject enrolled in the DIRECT Programme 8 June 2001 and last subject completed the DIRECT Programme 16 April 2008 mainly in hospital based clinics. 4514 patients type 1 diabetes were enrolled of whom 1421 proceeded to randomization, 711 to the candesartan arm and 710 to the placebo arm.
Pre-assignment Details: The most common reason for not being randomized was that all eligibility criteria were not fulfilled, followed by withdrawn informed consent.
Groups:
- Candesartan: Candesartan cilexetil 32 mg once daily
- Placebo: Placebo Comparator
Period: Overall Study
Arm/Group | Candesartan | Placebo
Started | 711 | 710
Completed | 605 | 618
Not Completed | 106 | 92
Not completed — Withdrawal by Subject | 73 | 67
Not completed — Death | 7 | 5
Not completed — Lost to Follow-up | 12 | 6
Not completed — Multiple Reasons | 14 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Candesartan | Placebo | Total
Number analyzed (Participants) | 711 | 710 | 1421
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.60 (8.0) | 29.90 (8.1) | 29.75 (8.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 298 | 318 | 616
  Male | 413 | 392 | 805

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a 2-step or Greater Increase in Early Treatment Diabetic Retinopathy Study (ETDRS) Severity Scale.
Description: Two steps were defined as either a 1-step change in each eye or as a 2-step change in one eye only. ETDRS is a scale with 11 steps (1-11, where a score of 1 represents no retinopathy and a score of 11 represents proliferative retinopathy). A generalized log-rank test was used to test difference between treatments.
Time Frame: From baseline to end of study, i.e. 5 years, with visits after a half year, one year and thereafter one visit per year.
Population: The population was the Intention To Treat population which includes all randomized patients with any post-randomization data.
Measure: Number; unit: Participants
Arm/Group | Candesartan | Placebo
Number analyzed (Participants) | 711 | 710
Participants | 178 (0.071) | 217 (0.086)
Statistical Analysis 1: Comparison: Candesartan vs Placebo; Test type: Superiority or Other; p = 0.0508, Log Rank; Generalized; Hazard Ratio (HR) = 0.821, 95% CI 2-sided [0.673 to 1.001]

2. Secondary Outcome: Rate of Change in Urinary Albumin Excretion Rate (UAER).
Description: An estimate of the slope from fitting a linear regression of log(UAER) over time for each patient.
Time Frame: From baseline to end of study, i.e. 5 years.
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: log (µg/min)/year
Arm/Group | Candesartan | Placebo
Number analyzed (Participants) | 711 | 710
log (µg/min)/year | 0.510 [0.487 to 0.534] | 0.543 [0.520 to 0.566]

ADVERSE EVENTS:
Time Frame: During treatment, up to 5 years.
Description: The population used was the safety population which includes all patients who received at least 1 dose of randomized study drug and for whom any post-randomization data were available.
Arm/Group | Candesartan | Placebo
Serious Adverse Events (participants affected / at risk) | 102/710 | 112/710
Other Adverse Events (participants affected / at risk) | 85/710 | 43/710
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Candesartan (N=710) | Placebo (N=710)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Bicytopenia (Blood and lymphatic system disorders) | 0 | 1
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 1 | 0
Lymphoid Tissue Hyperplasia (Blood and lymphatic system disorders) | 1 | 0
Myocardial Infarction (Cardiac disorders) | 0 | 4
Acute Coronary Syndrome (Cardiac disorders) | 0 | 1
Angina Pectoris (Cardiac disorders) | 1 | 0
Atrial Flutter (Cardiac disorders) | 0 | 1
Cardiac Failure Acute (Cardiac disorders) | 0 | 1
Coronary Artery Disease (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1
Pericardial Disease (Cardiac disorders) | 0 | 1
Pericardial Effusion (Cardiac disorders) | 0 | 1
Pericarditis (Cardiac disorders) | 0 | 1
Phimosis (Congenital, familial and genetic disorders) | 0 | 1
Basedow's Disease (Endocrine disorders) | 0 | 1
Hyperthyroidism (Endocrine disorders) | 1 | 0
Diplopia (Eye disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 2
Gastritis (Gastrointestinal disorders) | 1 | 2
Inguinal Hernia (Gastrointestinal disorders) | 0 | 2
Abdominal Pain (Gastrointestinal disorders) | 0 | 1
Appendicitis Perforated (Gastrointestinal disorders) | 1 | 0
Coeliac Disease (Gastrointestinal disorders) | 1 | 0
Colitis Ulcerative (Gastrointestinal disorders) | 0 | 1
Enteritis (Gastrointestinal disorders) | 1 | 0
Gastric Ulcer (Gastrointestinal disorders) | 1 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Haemorrhoidal Haemorrhage (Gastrointestinal disorders) | 1 | 1
Hiatus Hernia (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 1
Intestinal Obstruction (Gastrointestinal disorders) | 1 | 0
Mallory-Weiss Syndrome (Gastrointestinal disorders) | 0 | 1
Pancreatitis Chronic (Gastrointestinal disorders) | 0 | 1
Tooth Disorder (Gastrointestinal disorders) | 0 | 1
Chest Pain (General disorders) | 0 | 1
Generalised Oedema (General disorders) | 0 | 1
Cholecystitis Acute (Hepatobiliary disorders) | 0 | 1
Hepatitis (Hepatobiliary disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 2
Sarcoidosis (Immune system disorders) | 0 | 1
Gastroenteritis (Infections and infestations) | 9 | 1
Appendicitis (Infections and infestations) | 4 | 3
Pneumonia (Infections and infestations) | 3 | 2
Anogenital Warts (Infections and infestations) | 0 | 2
Bronchitis (Infections and infestations) | 2 | 0
Gastroenteritis Viral (Infections and infestations) | 1 | 2
Pharyngitis (Infections and infestations) | 2 | 0
Pilonidal Cyst (Infections and infestations) | 2 | 1
Pulmonary Tuberculosis (Infections and infestations) | 2 | 2
Pyelonephritis (Infections and infestations) | 2 | 0
Acute Sinusitis (Infections and infestations) | 1 | 0
Cat Scratch Disease (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 1 | 0
Gangrene (Infections and infestations) | 1 | 0
Hepatitis B (Infections and infestations) | 1 | 1
Hepatitis Viral (Infections and infestations) | 1 | 0
Pyelonephritis Chronic (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0
Tooth Abscess (Infections and infestations) | 0 | 1
Toxoplasmosis (Infections and infestations) | 0 | 1
Urinary Tract Infection (Infections and infestations) | 1 | 0
Viral Labyrinthitis (Infections and infestations) | 0 | 1
Viral Upper Respiratory Tract Infection (Infections and infestations) | 0 | 1
Ankle Fracture (Injury, poisoning and procedural complications) | 2 | 3
Facial Bones Fracture (Injury, poisoning and procedural complications) | 3 | 0
Hand Fracture (Injury, poisoning and procedural complications) | 0 | 2
Head Injury (Injury, poisoning and procedural complications) | 2 | 1
Multiple Injuries (Injury, poisoning and procedural complications) | 2 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 0 | 1
Foot Fracture (Injury, poisoning and procedural complications) | 0 | 1
Foreign Body In Eye (Injury, poisoning and procedural complications) | 0 | 1
Humerus Fracture (Injury, poisoning and procedural complications) | 0 | 1
Joint Dislocation (Injury, poisoning and procedural complications) | 1 | 0
Joint Injury (Injury, poisoning and procedural complications) | 0 | 1
Limb Crushing Injury (Injury, poisoning and procedural complications) | 1 | 0
Limb Injury (Injury, poisoning and procedural complications) | 1 | 0
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 1 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Road Traffic Accident (Injury, poisoning and procedural complications) | 1 | 1
Spinal Fracture (Injury, poisoning and procedural complications) | 1 | 0
Tendon Rupture (Injury, poisoning and procedural complications) | 1 | 0
Traumatic Amputation (Injury, poisoning and procedural complications) | 0 | 1
Blood Creatine Phosphokinase Increased (Investigations) | 0 | 1
HIV Test Positive (Investigations) | 1 | 0
International Normalised Ratio Increased (Investigations) | 0 | 1
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 12 | 17
Hypoglycaemia (Metabolism and nutrition disorders) | 17 | 16
Diabetes Mellitus Inadequate Control (Metabolism and nutrition disorders) | 1 | 6
Ketoacidosis (Metabolism and nutrition disorders) | 3 | 5
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 4
Dehydration (Metabolism and nutrition disorders) | 0 | 2
Hypoglycaemic Seizure (Metabolism and nutrition disorders) | 2 | 0
Shock Hypoglycaemic (Metabolism and nutrition disorders) | 1 | 0
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 2 | 2
Arthralgia (Vascular disorders) | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Compartment Syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Benign Neoplasm Of Thyroid Gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cervix Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Retroperitoneal Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Skin Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Teratoma Benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Thyroid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Convulsion (Nervous system disorders) | 1 | 2
Hypoglycaemic Coma (Nervous system disorders) | 2 | 2
Carpal Tunnel Syndrome (Nervous system disorders) | 0 | 1
Cerebral Infarction (Nervous system disorders) | 1 | 0
Cerebrovascular Accident (Nervous system disorders) | 1 | 1
Diabetic Autonomic Neuropathy (Nervous system disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 1 | 0
Guillain-Barre Syndrome (Nervous system disorders) | 1 | 0
Hydrocephalus (Nervous system disorders) | 0 | 1
Leukoencephalomyelitis (Nervous system disorders) | 0 | 1
Multiple Sclerosis (Nervous system disorders) | 1 | 1
Radiculitis Brachial (Nervous system disorders) | 1 | 0
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 2
Abortion (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Intra-Uterine Death (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Depression (Psychiatric disorders) | 3 | 1
Completed Suicide (Psychiatric disorders) | 0 | 1
Confusional State (Psychiatric disorders) | 1 | 0
Suicide Attempt (Psychiatric disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Ureteric Obstruction (Renal and urinary disorders) | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 0 | 2
Bartholin's Cyst (Reproductive system and breast disorders) | 0 | 1
Endometriosis (Reproductive system and breast disorders) | 1 | 0
Menstruation Irregular (Reproductive system and breast disorders) | 1 | 0
Ovarian Cyst (Reproductive system and breast disorders) | 0 | 1
Vaginal Haemorrhage (Reproductive system and breast disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal Polyps (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sleep Apnoea Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Skin Ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Candesartan (N=710) | Placebo (N=710)
Hypotension (Vascular disorders) | 85 | 43

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No